CLINICAL TRIAL: NCT01319188
Title: Ranibizumab for Age-Related Macular Degeneration and the Risk of Arterial Thromboembolic Events (RATE)
Brief Title: Ranibizumab and the Risk of Arterial Thromboembolic Events
Acronym: RATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated under the political pressure of the Federal Security Service of the Russian Federation (FSB) and the Russian Society of Cardiology
Sponsor: Ural State Medical University (Other)
Collaborators: Ural Institute of Cardiology (Other); De Haar Research Foundation (Other)
Responsible Party: Principal Investigator, Alexander Kharlamov, Scientific Assistant of C.E.O., Ural Institute of Cardiology, Ural State Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: RATE01
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Age-related Macular Degeneration; Coronary Artery Disease; Cerebrovascular Disorders
Keywords: Age-related macular degeneration; ranibizumab; acute thromboembolic events; coronary artery disease; cerebrovascular disease
MeSH Terms: conditions — Macular Degeneration; Coronary Artery Disease; Cerebrovascular Disorders | interventions — Ranibizumab; Photochemotherapy; Laser Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.5 mg of ranibizumab (Active Comparator)
  Interventions: Drug: 0.5 mg of ranibizumab
- injection + photodynamic therapy (Active Comparator)
  Interventions: Procedure: 0.5 mg of ranibizumab + photodynamic therapy
- Sham injection (Sham Comparator)
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: 0.5 mg of ranibizumab — Intravitreous ranibizumab (0.5 mg, injections at four week intervals for six months followed by further treatment at three month intervals with total duration of treatment until 24 months).
  Other Names: Lucentis
  Arms: 0.5 mg of ranibizumab
Procedure: 0.5 mg of ranibizumab + photodynamic therapy — Photodynamic treatment with ranibizumab for predominantly classic type neovascular age related macular degeneration.
  Other Names: Lucentis + laser therapy
  Arms: injection + photodynamic therapy
Other: Sham injection — Sham treatment for occult or minimally classic type neovascular age related macular degeneration.
  Other Names: Sham comparator
  Arms: Sham injection

SUMMARY:
The investigators assume that ranibizumab might be dangerous in patients with history of coronary artery disease or cerebrovascular events. The main objective of study is to reveal contraindications for ranibizumab prescription in patients with history of coronary artery disease and cerebrovascular events. Moreover, an association between management with ranibizumab and ATE rate in healthy above 50 years old persons is a concern of great interest as well.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a degenerative condition affecting the macula or central area of the retina in elderly people. Early AMD is marked by the presence of soft drusen and/or retinal pigment abnormality (hyper- and hypopigmentation). Late AMD includes 2 forms, nonneovascular (dry) AMD and neovascular (wet) AMD. Despite new medical and surgical interventions, AMD remains a leading cause of vision loss in elderly people all over the world.

Ranibizumab is one of the most effective approaches of AMD management. Ranibizumab - a recombinant, humanized, monoclonal antibody Fab that neutralizes all active forms of vascular endothelial growth factor A (VEGF A) - has been evaluated for the treatment of AMD. Ranibizumab binds to the receptor binding site of active forms of VEGF-A. VEGF-A cause neovascularization and leakage in models of ocular angiogenesis and vascular occlusion, and is thought to contribute to the progression of neovascular AMD and macular edema following RVO. Prevents the interaction of VEGF-A with its receptors (VEGFR1 and VEGFR2) on the surface of endothelial cells, reducing endothelial cell proliferation, vascular leakage, and new blood vessel formation.

There have been a number of studies that have examined a possible association between ranibizumab and arterial thromboembolic events (ATE). The ATE rate in the three controlled neovascular AMD studies during the first year was 1.9% (17 out of 874; 0.3-0.5 mg LUCENTIS) vs 1.1% (5 out of 441) in control arms (AMD-1, AMD-2). In the second year the ATE rate was 2.6% (1323 patients; Lucentis 879) vs Control 444 (p < 0.05). The ATE rate in the two controlled RVO studies (RVO-1, RVO-2) during the first six months was 0.8% (789 patients; Lucentis 527 vs Sham 262).

The investigators assume that ranibizumab can be rather dangerous in patients with history of coronary artery disease or cerebrovascular events. The main objective of study is to reveal contraindications for ranibizumab prescription in patients with history of coronary artery disease and cerebrovascular events. Moreover, an association between management with ranibizumab and ATE rate in healthy above 50 years old persons is a concern of great interest as well.

ELIGIBILITY:
Inclusion Criteria:

* age - 50 years old and older
* male and female
* age-related macular degeneration (AMD)
* have a lesion in the study eye with a total size of less than 12 optic disc areas for minimally classic or occult lesions but no more than 5400 μm in greatest linear dimension for predominantly classic lesions
* have best corrected visual acuity of 6/12 to approximately 6/96 (Snellen equivalent), assessed with the use of charts from the Early Treatment Diabetic Retinopathy Study (ETDRS) (70 to 25 ETDRS 1 m equivalent letter scores; patients initially view the charts at a starting distance of 4 m, the number of correctly read letters are given a correction factor with the final letter score being the equivalent of a patient reading it at 1m. A score of 55 letters approximates to 6/24 Snellen acuity)
* have no permanent structural damage to the central fovea
* have had no previous treatment for exudative age related macular degeneration
* healthy subjects (no history of cardio- or cerebrovascular events), or history of coronary artery disease (cardiovascular events - myocardial infarction, unstable angina), or history of cerebrovascular events (brain ischemia, and/or stroke), but not in the preceding six months

Exclusion Criteria:

* history of cardiovascular events (myocardial infarction, unstable angina) or cerebrovascular events in the preceding six months
* stenting, or any surgery in the preceding six months
* other acute illnesses in the preceding three months
* III-IV NYHA functional class of heart failure
* mental and brain disorders
* pregnancy
* family hypercholesterolemia
* blood disorders
* malignant tumors
* participation to any drug investigation during the previous three months

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Arterial thromboembolic events rate | at month 6, 12 and 24
  This is a combined primary outcome that included:
  * all cause mortality
  * nonfatal stroke
  * nonfatal myocardial infarction
  * vascular death

SECONDARY OUTCOMES:
Serum concentration of ranibizumab | at month 6, 12 and 24
  Serum concentration of ranibizumab
Serum VEGF | at month 6, 12 and 24
  Measurement of serum VEGF
Mean change in visual acuity (letters) | at month 6, 12 an 24
  mean change in visual acuity (letters)
Coronary and/or cerebral stenting, and/or CABG rate | at month 6, 12 an 24
  Coronary and/or cerebral stenting, and/or CABG rate
Total cholesterol | at month 6, 12 and 24
  Total cholesterol measurement
Systolic blood pressure | at month 6, 12 and 24
  Systolic blood pressure
NYHA (New York Heart Association) functional class of heart failure | at month 6, 12 and 24
  NYHA (New York Heart Association) functional class of heart failure
Diabetes mellitus morbidity | at month 6, 12 and 24
  Diabetes mellitus morbidity
Serum fibrinogen | at month 6, 12 and 24
  Serum fibrinogen measurements
Serum C-RP | at month 6, 12 and 24
  Serum C-RP measurements
Serum D-dimer | at month 6, 12 and 24
  Serum D-dimer measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gabinsky, M.D., Ph.D., Study Chair — Ural Institute of Cardiology; Alexander Kharlamov, M.D., Ph.D., Study Director — Ural State Medical University; Olga Kovtun, M.D., Ph.D., Principal Investigator — Ural State Medical University
Locations (2):
- De Haar Research Foundation, Rotterdam, South Holland, Netherlands
- Ural Institute of Cardiology, Yekaterinburg, Russia

REFERENCES:
- See also: Ural Institute of Cardiology — http://www.cardio-burg.ru